CLINICAL TRIAL: NCT01636895
Title: An Evaluation of Sulfadoxine-pyrimethamine Resistance and Effectiveness of IPTp in Nigeria
Brief Title: Evaluation of SP Resistance and Effectiveness of IPTp in Nigeria
Acronym: OR1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaria Consortium, UK (Network)
Collaborators: Department for International Development, United Kingdom (Other Government); London School of Hygiene and Tropical Medicine (Other); University of Nigeria, Enugu Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SuNMaP-OR1
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy Complications Parasitic
Keywords: malaria; pregnancy; prevention; treatment; molecular markers
MeSH Terms: conditions — Pregnancy Complications, Parasitic; Malaria | interventions — Pyrimethamine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SP-IPTp efficacy (Experimental): Efficacy of suphladoxine/pyrimethamine as IPTp
  Interventions: Drug: Efficacy of suphladoxine/pyrimethamine as IPTp

INTERVENTIONS:
Drug: Efficacy of suphladoxine/pyrimethamine as IPTp — 3 tablets (single dose)given twice during pregnancy one month apart after quickening
  Other Names: Fansidar
Drug: Efficacy of suphladoxine/pyrimethamine as IPTp — 2 courses of 3 tablets of 500 mg N1-(5,6-dimethoxy-4-pyrimidinyl) sulfanilamide (sulfadoxine) and 25 mg 2,4-diamino-5-(p-chlorophenyl)-6-ethylpyrimidine (pyrimethamine)administered (at least 1 month apart) as DOTs to pregnant mother after quickening
  Other Names: Fansidar

SUMMARY:
The study has two components: component A is a cohort study to determine the in vivo efficacy of SP to clear and prevent malaria parasitaemia in asymptomatic pregnant women and component B is a cross sectional study of women delivering at the study hospitals to assess the effectiveness of SP-IPTp to reduce adverse maternal and birth outcomes in the current context of increasing SP resistance. Results of component A and B studies will be used to model the relationship between the prevalence of molecular markers of SP resistance, in vivo efficacy to clear parasite and the effectiveness of SP-IPTp and to develop guidelines for routine monitoring effectiveness of SP-IPTp as part of ANC surveillance.

DETAILED DESCRIPTION:
Study sites will include different levels of transmission and social factors affecting ANC attendance Damboa hospital in Borno state has a catchment area with pop of 231,573 with a semi arid climate and where malaria is mesoendemic. The expected number of patients is 15-25 per week for new bookings Park Lane hospital serves a semiurban population. Malaria transmission is holoendemic and stable. 1400 women attend ANC services per month Women will receive SP-IPTp according to National guidelines and will be followed for 42 days to assess the therapeutic efficacy in parasitaemic women and to assess the ability to remain parasite free. PCR will be used to determine reinfection from recrudescence

ELIGIBILITY:
Inclusion Criteria:

* gestational age 16-30 weeks
* Axillary temperature ,37.5 Degrees
* informed consent

Exclusion Criteria:

* gravida > 2
* previous inclusion in this study
* history of hypersensitivity to SP or components of SP
* Use of IPTp with SP during this pregnancy
* history of taking other antimalarials in the past month
* Known HIV infection

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of SP-IPTp for clearing peripheral malaria parasiteamia in asymptomatic primi and secondi gravid women | 15 months
  PCR corrected Adequate parasitological clearance by day 42

SECONDARY OUTCOMES:
To determine the efficacy of SP-IPTp in preventing new infections in primi- and secundi-gravid women | 15 months
  PCR uncorrected parasitological clearance by day 42
To estimate the prevalence of molecular markers of SP resistance in primi- and secundi-gravid women | 15 months
  Prevalence of molecular markers of SP resistance at enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chandramohan, PHD, Study Chair — London School of hygeine and tropical medicine; Elvis N Shu, PHD, Principal Investigator — College of Medicine, University of Nigeria , Enugu Campus; Ebenezer S Baba, MBBS, MPH, Study Director — Malaria Consortium
Locations (1):
- Damboa Hospital Borno state and Park Lane hospital Enugu state, Enugu, Borno State and Enugu State, Nigeria